CLINICAL TRIAL: NCT00550472
Title: Intervention Study on the Effects of a Probiotic Yoghurt Drink on the Immune System and Further Physiological Parameters in Patients With Atopic Dermatitis and Healthy Persons
Brief Title: The Effect of a Probiotic Intervention in Healthy Subjects and Patients With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: University of Jena, Dept. of Nutritional Physiology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LSEP H18-05
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Atopic Dermatitis
Keywords: probiotics; atopic dermatitis; immune system; human; Lactobacillus; Bifidobacterium; healthy subjects
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probiotic (Experimental): intervention
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — Lactobacillus paracasei Lpc-37, Lactobacillus acidophilus 74-2 Bifidobacterium animalis subsp. lactis DGCC 420

SUMMARY:
The study was performed to investigate the effects of a probiotic supplementation containing Lactobacillus paracasei Lpc-37, Lactobacillus acidophilus 74-2 and Bifidobacterium animalis subsp. lactis DGCC 420 (B. lactis 420) on clinical, immunological and faecal parameters in healthy volunteers and in patients with atopic dermatitis (AD).

DETAILED DESCRIPTION:
Recent studies suggest that oral bacteriotheraphy with probiotic bacteria might be useful to alleviate atopic dermatitis in infants. There are few indications about the effect of probiotics in the management of atopic dermatitis in adults.

As a precondition for participating in this study, the subjects were provided information in writing and verbally about the details of the study. Informed consent was obtained from all volunteers. Before the beginning of the study, all participants were subject to a medical examination in the Clinic for Dermatology and Dermatologic Allergology of the Friedrich Schiller University Jena. The AD was diagnosed according to the atopy-score of Diepgen. Severity of eczema was evaluated by using the SCORAD score. A skin prick test was performed for the exclusion of type 1 sensitivity to cow's milk.

The study was designed as a placebo-controlled and cross-over study. After a 3-week run-in period the 30 participants (15 healthy subjects and 15 patients with AD) were randomized to receive either 200 ml/d of a probiotic drink containing L. paracasei Lpc-37, L. acidophilus 74-2 and B. lactis 420 or 200 ml/d of a placebo drink for 8 weeks. After a 2-week washout period the intervention was crossed between the groups and the respective products were consumed for another 8 weeks followed by a 2-week washout period. Venous blood and fresh stool samples were collected before the beginning and at the end of each period. In AD patients the Scoring of atopic dermatitis (SCORAD) was assessed by the same physician every 4 weeks and 2 weeks after the wash-out period, respectively.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* No allergic asthma
* No allergic rhinoconjunctivitis
* No food allergies
* Exclusion of atopic diathesis (< 7 points in Erlangen atopy score)

Patients with AD:

* Clear diagnosis of atopic dermatitis (> 10 points in the Erlangen atopy score) or flexural eczema or pruritis for at least 12 months (recidivating or permanent)
* SCORAD 5-30 (minor or medium AD)
* Willingness to apply for the duration of the study exclusively the cosmetic products recommended by the accompanying doctor and to use the recommended class II corticosteroid (Advantan) as further therapy of AD (for example during an episode)

Exclusion Criteria:

* Pregnancy, lactation
* Immune suppressive or cytostatic therapy or systemic steroids < 1 month before the first intake
* Phototherapy or systemic therapy of AD < 1 month before the first intake
* Active infections of the skin
* Relevant asthma disease, which must be treated with inhalative corticoids (FEV1 < 70 %)
* Patients with an indigestibility of/allergy against the components of milk/lactose intolerance (previously known or detected in the allergy test)
* Patients under long-term treatment with systemic steroids, depot steroids, long-acting antihistamines, tranquilizers, psychopharmaceuticals
* Intake of antihistamines, psychopharmaceuticals with antihistaminic effect and application of steroid containing cream to the forearms within the past 7 days before prick testing resp. treatment of the patient with Astemizol (Hismanal) within 4 weeks before the test. Such patients must be excluded from the study because of the long half-life of the medicament.
* Acute or chronic symptomatic heart disease or severe internistic diseases
* Autoimmune diseases, immune deficiencies (including immune suppressive treatment)
* Immune-complex-induced immunopathies or malignant tumors
* Abuse of alcohol, drugs or medicaments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
SCORAD change in patients with AD taken at baseline and after 4 and 8 weeks, respectively -change in phagocytic and oxidative burst activity of monocytes and granulocytes at baseline and after 8 weeks | 8 weeks

SECONDARY OUTCOMES:
cellular and humoral immunological parameters (CD's; Interleukins); detection of bacterial species in faecs, faecal short-chain fatty acids, blood lipids | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — University of Jena, Dept. of Nutritional Physiology
Locations (1):
- University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Thuringia, Germany